CLINICAL TRIAL: NCT00848991
Title: Comparison of Propofol Standard Anesthetic to Precedex With Propofol for Emergence and Recovery in Patients Having Craniotomy Surgery
Brief Title: Comparison of Propofol to Precedex With Propofol for Emergence and Recovery in Patients Having Craniotomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Dr. Michael Misbin, Cooper University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2008-12-17; First posted 2009-02-23 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Cranitomy Surgery
Keywords: precedex; propofol
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precedex (Active Comparator): In the operating room routine anesthesia monitors will be placed and vital signs will be recorded continuously using data collection software. A routine propofol anesthetic will be administered to subjects randomized to the control group or a Precedex infusion with propofol for subjects randomized to the treatment group. Precedex infusion will be started after induction of general anesthesia. Vital signs (SBP, DBP, MAP) will be recorded continuously throughout the surgery. At the end of the case subjects will be extubated and the blinded observer will assess emergence from anesthesia based on hemodynamic stability and tolerance of the endotracheal tube. Videotaping of emergence will be used to assist in the evaluation of emergence of anesthesia and extubation.
  Interventions: Drug: Precedex
- Propofol (Active Comparator): Propofol for emergence from anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Precedex — Subjects randomized to the comparison group will receive a standardized general anesthetic. Anesthesia will be induced with propofol 1.5 ? 2.5 mg/kg, rocuronium 0.6 mg/kg, and sufentanil 0.1 ? 1mcg/kg. Anesthesia will be maintained with an infusion with propofol 25 -200 mcg/kg/min, sufentanil 0.0025 - 0.03 mcg/kg/min, and zemuron as needed. For the Precedex group the drug will be infused at 0.3-0.7 mcg/kg/hr. Blood pressure will be maintained within 10% of baseline prior to opening of the dura, subsequently to be maintained between a systolic of 100 ? 130 mmHg. Hypertension will be managed with standardized amounts of labetalol and nicardipine. Morphine will be titrated as needed to a maximum of 0.05mcg/kg at the conclusion of case. Hemodynamic data and emergence evaluations will be collected in the operating room, pre-induction until the end of anesthesia and discharge from the operating room. There will be no further follow up.
  Arms: Precedex
Drug: Propofol — evaulation of propofol for emergence from anesthesia
  Arms: Propofol

SUMMARY:
Primary Hypothesis: The use of a Precedex infusion, in addition to propofol during surgery, will improve patient management through the anesthesia postoperative recovery period determined by improvement in patients? tolerance of the endotracheal tube.

Secondary hypothesis: The use of a Precedex infusion, in addition to propofol during surgery will provide improved hemodynamic stability.

DETAILED DESCRIPTION:
The purpose of this study is to compare the addition of Precedex to a propofol intravenous anesthetic for emergence from anesthesia in patients having craniotomy surgery for brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1, 2, and 3

Exclusion Criteria:

* ASA status 4 and 5 patients
* Patients with positive pregnancy tests

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The use of Precedex for craniotomy surgery offers the potential for improved hemodynamic control and improved tolerance of the endotracheal tube, therefore potentially benefiting these patients. | 4 hours after awaking from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Misbin, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States